CLINICAL TRIAL: NCT02776475
Title: Are the Effects of Sacral Neuromodulation for Urinary Urgency, Frequency, and Urge Incontinence Maintained With the Device Temporarily Turned Off?
Brief Title: The Effects of Sacral Neuromodulation for Urinary Urgency, Frequency, and Urge Incontinence
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficult to find eligible patients for enrolling
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-019
Record Dates: First submitted 2016-05-03; First posted 2016-05-18 (Estimated); Last update posted 2022-11-10 (Actual); Status verified 2020-10

CONDITIONS: Urinary Urge Incontinence
MeSH Terms: conditions — Urinary Incontinence, Urge

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sacral neuromodulation device turned off (Other): Patients who are currently being successfully treated with sacral neuromodulation for the primary diagnosis of urinary urge incontinence or urgency and frequency (implantation for minimum 12 months) will be to have the sacral neuromodulation device turned off for four consecutive weeks.
  Interventions: Procedure: Sacral neuromodulation device turned off

INTERVENTIONS:
Procedure: Sacral neuromodulation device turned off — Each patient will be to have the sacral neuromodulation device turned off for four consecutive weeks.

SUMMARY:
This prospective one group cohort study seeks to investigate the effects of sacral neuromodulation on urinary urgency, frequency and urge incontinence are maintained after the simulator device is temporarily turned off for a period of four weeks.

DETAILED DESCRIPTION:
Urinary urgency, frequency, and urge incontinence are very common symptoms, affecting up to one in three adults in the United States. The total economic cost of these disorders was estimated to be above $12 billion in the year 2000, with the vast majority being for women.

Sacral neuromodulation (SNM) has become a popular and successful treatment option for people who suffer from these conditions. Sacral neuromodulation device delivers electrical pulses to an area near the sacral nerve.

There has been some data published which showed that for patients with fecal incontinence, symptom relief can persist for significant time periods despite having the stimulator device turned off. Based on their findings, potential exists to prolong battery life if patients can cycle the on and off periods for their device while keeping their symptoms stable.

The typical battery life of the implantable pulse generator (IPG) is approximately 5 years depending on the system settings. When the IPG is at the end of its battery life, a new IPG must be implanted. The cost of replacing the IPG ranges from $13,952 to $16,470. IPG replacement must be done in the operating room and requires the patient to undergo anesthesia and its associated risks.

This study will investigate whether the symptoms of urinary urgency, frequency, and urge incontinence remain stable in patients with SNM with the device turned off for a period of four weeks.

Current Cincinnati Urogynecology Associates (CUA) patients who are currently being successfully treated with sacral neuromodulation for the primary diagnosis of urinary urge incontinence or urgency and frequency who elect participate in the study will have the device turned off for four consecutive weeks. Their symptoms will be monitored during this time period.

ELIGIBILITY:
Inclusion Criteria:

* Women, aged 18-85 with who have previously had the InterStim device implanted and have experienced good control of their symptoms for at least one year.

Exclusion Criteria:

* Patients with less than 6 months of expected battery life on their device established at office testing.
* Patients with poor control of their symptoms within the last one year.
* Patients with degenerative neurological disorders or spinal cord injuries.
* Patients with cognitive disabilities or those lacking the mental capacity to understand and answer questionnaires.
* Patients who are pregnant or may become pregnant.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-08-04 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
The difference in scores on the International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF) from baseline with the SNM device compared to having the device turned off for a period of four weeks | The outcome measure is assessing change between initial baseline and 4 weeks after turning off the device.
The difference in scores on the International Consultation on ICIQ-SF from baseline with the SNM device compared to having the device turned off for a period of up to six months | The outcome measure is assessing change between initial baseline and 6 months after turning off the device.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Pauls, MD, Principal Investigator — TriHealth - Cincinnati Urogynecology Associates
Locations (1):
- Cincinnati Urogynecology Associates, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No